CLINICAL TRIAL: NCT05936593
Title: Migration in a Cruciate Retaining and a Condylar Stabilizing Insert of a Robot-assisted Uncemented Total Knee Prosthesis Using Model-based RSA: a Mono-Center Randomized Controlled Trial With 10 Years Follow-up
Brief Title: Migration of CS vs CR Insert in TKA Using RSA
Acronym: CS vs CR RSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OC-2021-004
Record Dates: First submitted 2023-06-12; First posted 2023-07-10 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Wear of Articular Bearing Surface of Prosthetic Joint; Migration of Implant
Keywords: Total knee arthroplasty; Insert
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Condylar Stabilizing (CS) insert (Active Comparator)
  Interventions: Device: Condylar Stabilizing (CS) insert
- Cruciate Retaining (CR) insert (Active Comparator)
  Interventions: Device: Cruciate Retaining (CR) insert

INTERVENTIONS:
Device: Condylar Stabilizing (CS) insert — During TKA surgery a Condylar Stabilizing (CS) insert is implanted and tantalum beads are placed around the prosthesis.
  Arms: Condylar Stabilizing (CS) insert
Device: Cruciate Retaining (CR) insert — During TKA surgery a Cruciate Retaining (CR) insert is implanted and tantalum beads are placed around the prosthesis.
  Arms: Cruciate Retaining (CR) insert

SUMMARY:
Background:

The choice whether or not to preserve the posterior cruciate ligament (PCL) in total knee arthroplasty (TKA) is coupled to the us of a PCL-retaining (CR) or a condylar (CS) insert. The CS insert is anterior-lipped (AL) to prevent anterior translation of the femur on the tibia with flexion and compensate the function of the PCL. Currently both the CR and CS insert are made of highly cross-linked polyethylene (HXPLE) to theoretically reduce wear related osteolysis. However, this also might diminish the fracture toughness and crack propagation of the insert. The investigators expect that due to the high contact forces on the anterior lip of the CS insert during flexion, especially in younger and more active patients, and the lower fracture toughness of HXPLE, the CS insert insert might show more migration, wear or other damage compared to the CR insert in the long-term, which might lead to more revisions in the CS insert compared to the CR insert.

To measure the migration and wear, during surgery tantalum markers will be inserted in the host bone using a marker inserter. The displacement of the prosthesis with reference to the host bone will be measured using model-based RSA. Both tantalum markers ande the inserter are already used for study purposes. However, the safety and usability are not registered before.

Objective:

The primary objective is to compare the migration of both the femoral and tibial component by the use of a CS insert or CR insert both made of HXPLE using model-based roentgen stereophotogrammetric analysis (mRSA). Furthermore, the safety and usability of the tantalum markers and the marker inserter will be determined. The secondary objective is to determine the influence of the type of insert on the wear, inducible displacement, survival and clinical outcomes.

Study design:

A randomized controlled trial

Study population:

Forty-four patients scheduled to undergo primary total knee replacement, aged below 70 years with an ASA-score of 1 or 2 will be needed in total, divided in two groups of 22 patients each.

Intervention:

One group receives an uncemented TKP with a CS insert, while the other group receives an uncemented TKP with a CR insert. Both will be placed using the MAKO-robotic arm using a kinematic balancing technique.

Outcomes:

Main study parameters are migration of the femoral and tibial components measured with model-based RSA software till 10 years postoperatively. Furthermore, the stability of the markers will be determined and the complications due to the markers and/or the marker inserter will be registered. The secondary parameters are wear, inducible displacement, survival, clinical outcomes and complications up to 10 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo primary total knee replacement with the MAKO-robotic arm, with one of the following indications:
* Painful, disabling joint disease of the knee resulting from: non-inflammatory degenerative joint disease (including osteoarthritis, traumatic arthritis or avascular necrosis) or rheumatoid arthritis.
* One or more compartments are involved;
* Moderate varus, valgus, or flexion deformity in which the ligamentous structures can be returned to adequate function and stability (meaning a varus, valgus or flexion deformity < 15 degrees);
* Age between 18 and 70 years;
* ASA score I or II;
* A good nutritional state of the patient;
* Patients with a completely intact PCL at the time of surgery;
* Patient is able to understand the study and is willing to participate and to sign the Informed Consent;
* Patient is able to speak and write Dutch.

Exclusion Criteria:

* Contraindications manufacturer:
* Any active or suspected latent infection in or about the knee joint;
* Distant foci of infection which may cause hematogenous spread to the implant site;
* Any mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in postoperative care;
* Bone stock compromised by disease, infection or prior implantation which cannot provide adequate support and/or fixation to the prosthesis;
* Skeletal immaturity;
* Severe instability of the knee joint secondary to the absence of collateral ligament integrity and function;
* Metal in the operative or non-operative leg which lead to the creation of accuracy-reducing artefacts in the CT scan;
* Body Mass Index (BMI) of > 35 kg/m2;
* Flexion contracture of 15 degrees and more;
* Varus/valgus contracture of 15 degrees and more;
* History of total or unicompartmental reconstruction of the affected joint;
* Bilateral operation;
* A Total Hip Arthroplasty (THA) on contralateral and/or ipsilateral side within the last year that is considered to have an unsatisfactory outcome (Patients with contralateral and/or ipsilateral THA > 1 year ago with good outcome can be included in the study);
* A Total Knee Arthroplasty (TKA) on contralateral side within the last 6 months that is considered to have an unsatisfactory outcome. (Patients with contralateral TKA > 6 months ago with good outcome can be included in the study);
* Patients who will need lower limb joint replacement for another joint within one year.
* Active or suspected latent infection in or about the knee joint;
* Osteomyelitis;
* Sepsis;
* A systemic or metabolic disorder leading to progressive bone deterioration, excluding rheumatoid arthritis;
* Vascular insufficiency, muscular atrophy;
* Neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device;
* Female patients planning a pregnancy during the course of the study;
* The patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements.
* Patients bone stock is compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis;
* A knee fusion to the affected joint;
* Patient has a known or suspected sensitivity or allergy to one or more of the implant materials;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Translations (mm) | 10 years after surgery
  The translations of the femoral and tibial components measured in 3 axis (z, y and z) with model-based RSA over 10 years.
Rotations (degrees) | 10 years after surgery
  The rotations of the femoral and tibial components measured in 3 axis (z, y and z) with model-based RSA over 10 years.
Stability of the tantalum markers | 10 years after surgery
  Stability of the tantalum markers will be determined by the mean error value of the markers.
Safety of the tantalum markers and the inserter | 10 years after surgery
  Safety of the tantalum markers are determined by registration of the complications due to the markers and/or marker inserter. Complications will be expressed by numbers and percentages.

SECONDARY OUTCOMES:
Wear | 10 years after surgery
  Wear of the insert measures in 3 axis (x, y and z)
Inducible displacement (mm) | 10 years after surgery
  The inducible displacement gives insight into the nature and durability of the fixation and is defined as the micromotion occurring in response to external forces. The inducible displacement will be expressed by translations (x-, y- and z-direction) in mm
Inducible displacement (degrees) | 10 years after surgery
  The inducible displacement gives insight into the nature and durability of the fixation and is defined as the micromotion occurring in response to external forces. The inducible displacement will be expressed by rotations (x-, y- and z-direction) in degrees.
Survival | 10 years after surgery
  Survival of the CS and CR inserts is measured by registration of all complications and is expressed by numbers and percentages.
Clinical outcomes: Knee Society Score (KSS) | 10 years after surgery
  The Knee Society Score (KSS) is a questionnaire to rate the knee prosthesis function. A high score means a good function and a low score means a worse function. The score varies between 0 and 100.
Clinical outcomes: Numeric Rating Scale for pain (NRS pain) | 10 years after surgery
  The Numeric Pain Rating Scale (NRS) measures the amount of pain experienced in the past week during rest and activity. It is a scale from 0 (no pain) to 10 (worst pain imaginable)
Clinical outcomes: EuroQol 5D (EQ-5D-5L) | 10 years after surgery
  The EuroQol-5D-5L (EQ-5D-5L) is a questionnaire that describes the overall health condition of the person. The score is given by an index consisting of 5 numbers, which represents a health status. A lower score indicates a good condition. The last question of this questionnaire is the overall health condition of the person on a scale of 0 to 100. In this question a higher score indicates a good condition.
Clinical outcomes: Knee Injury and Osteoarthritis Outcome Score (short version, KOOS-PS) | 10 years after surgery
  The Knee Injury and Osteoarthritis Outcome Score - short version (KOOS-PS) is a questionnaire about the ability to perform normal daily activities. A high score means that the activities cost a lot of effort to perform, while a low score means that the activities can be done with minimum effort. The score varies between 0 and 100.
Clinical outcomes: Forgotten Joint Score (FJS) | 10 years after surgery
  The Forgotten Joint score (FJS) is a questionnaire about the awareness of the prosthetic knee. A high score means a low awareness and a low score means a high awareness. The score varies between 0 and 100.
Clinical outcomes: Numeric Rating Scale for Satisfaction (NRS satisfaction) | 10 years after surgery
  The satisfaction is a single question about the overall satisfaction of the result of the surgery on a scale from 0 (very unsatisfied) to 10 (very satisfied).
Clinical outcomes: Oxford Knee Score (OKS) | 10 years after surgery
  The Oxford Knee Score (OKS) is a questionnaire about the amount of influence of the operated knee on the persons life. A low score means that the life of the person is influenced a lot by the operated knee, while a high score means that the life of the persons is little influenced by the operated knee. The score varies between 0 and 48.

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier Haga Orthopedisch Centrum, Zoetermeer, South Holland, Netherlands